CLINICAL TRIAL: NCT05131854
Title: Incidence , Risk Factors and Outcomes of Haemodynamic Instability and Cardiac Arrest During Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Essamedin Mamdouh Negm, principal investigator, Zagazig University
Other Study IDs: 8078-13-10-2021
Record Dates: First submitted 2021-10-15; First posted 2021-11-23 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Spine Surgery
Keywords: spine surgery , bradycardia , cardiac arrest
MeSH Terms: conditions — Bradycardia; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Risk factors for cardiac arrest during spine surgery have been well defined, including lumbar fusion, age over 65 years, obesity, cardiovascular disease, ethnicity and ASA status. Bradycardia and asystole have been described under general anaesthesia in combined surgical cohorts: Proposed mechanisms include unopposed parasympathetic activation, enhanced vasovagal response to decreased venous return, and psychiatric stressors. The investigators prospectively will review patients candidates for spine surgery to explore potential incidence, contributory factors and outcomes to unexpected transient intraoperative haemodynamic instability, arrhythmia, and cardiac arrest during spine surgery as these data are needed to aid risk stratification and improve decision making for spine care teams.

ELIGIBILITY:
Inclusion Criteria:

1. Aged more than 18
2. Gender: both.
3. ASA grade I-II (American society of anesthiologists).
4. Prepared to spine surgery under general anesthesia

Exclusion Criteria:

1. Ischemic heart patients
2. Hypertensive patients
3. Patients with atrial fibrillation or any previous history of attack of arrhythmias
4. Patients on B.B ( beta-blockers)
5. Chronic use of neuropsychiatric medications
6. Renal Impairment
7. Liver Dysfunction.
8. Any complications during the procedure as massive hemorrhage
9. Surgery for traumatic spinal cord

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: population candidated for spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Haemodynamic Instability during Spine Surgery | allover one year
  To calculate Incidence of Haemodynamic Instability during Spine Surgery
Risk factors of Haemodynamic Instability during Spine Surgery | allover one year
  To analyze risk factors of Haemodynamic Instability during Spine Surgery
outcomes of Haemodynamic Instability during Spine Surgery | allover one year
  To calculate the rate of mortality of Haemodynamic Instability during Spine Surgery
Incidence of cardiac arrest during Spine Surgery | allover one year
  To calculate Incidence of cardiac arrest during Spine Surgery
Risk factors of cardiac arrest during Spine Surgery | allover one year
  To analyze risk factors of cardiac arrest during Spine Surgery
outcomes of Cardiac Arrest during Spine Surgery | allover one year
  To calculate the rate of mortality of cardiac arrest during Spine Surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Egypt